CLINICAL TRIAL: NCT01713270
Title: Safety and Effectiveness Study of Percutaneous Catheter-based Renal Sympathetic Denervation in Patients With Drug-resistant Hypertension and Symptomatic Atrial Fibrillation
Brief Title: Renal Sympathetic Denervation in Patients With Drug-resistant Hypertension and Symptomatic Atrial Fibrillation
Acronym: RSDforAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Qijun Shan, Professor，Director, Cardiac Arrhythmia Group, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-SR-080
Record Dates: First submitted 2012-10-18; First posted 2012-10-24 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-07

CONDITIONS: Hypertension; Atrial Fibrillation
Keywords: Hypertension; Atrial Fibrillation; Arrhythmias, Cardiac; Heart Diseases
MeSH Terms: conditions — Hypertension; Atrial Fibrillation; Arrhythmias, Cardiac; Heart Diseases | interventions — Pharmaceutical Preparations; Electric Countershock

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- renal sympathetic denervation (Experimental): Contrast renal angiography was performed to localize and assess the renal arteries. Once the anatomy was deemed acceptable, the internally irrigated radiofrequency ablation catheter was introduced into each renal artery. This was then maneuvered within the renal artery to allow energy delivery in a circumferential, longitudinally staggered manner to minimize the chance of renal artery stenosis. About four to eight ablations at 10 W for 60 seconds each were performed in both renal arteries. After renal sympathetic denervation, patients with persistent AF accepted direct-current cardioversion immediately.
  Interventions: Procedure: renal sympathetic denervation; Drug: drug; Procedure: Direct-Current Cardioversion
- drug therapy (Active Comparator): Patients in the drug treatment group will be followed-up at 3, 6, 9 and 12 months after randomization. All the patients in this group will take their baseline antihypertensive medication at the original doses, without any changes except when medically required. Antiarrhythmic drugs treatment is consistent in both arms.
  Interventions: Drug: drug

INTERVENTIONS:
Procedure: renal sympathetic denervation — Contrast renal angiography was performed to localize and assess the renal arteries for accessibility and appropriateness for RSD. Once the anatomy was deemed acceptable, the internally irrigated radiofrequency ablation catheter(Celsius Thermocool, Biosense Webster, Diamond Bar, California) was introduced into each renal artery. then was maneuvered within the renal artery to allow energy delivery in a circumferential, longitudinally staggered manner to minimize the chance of renal artery stenosis. About four to eight ablations at 10 W for 1 minute each were performed in both renal arteries. During ablation, the catheter system monitored tip temperature and impedance, altering radiofrequency energy delivery in response to a predetermined algorithm.
  Other Names: renal denervation; renal ablation
  Arms: renal sympathetic denervation
Drug: drug — Angiotensin converting enzyme inhibitors, angiotensin receptor antagonist, calcium antagonists, diuretic, beta adrenoceptor blocking agents, propafenone, amiodarone
Procedure: Direct-Current Cardioversion — After renal sympathetic denervation, Persistent AF individual (except intracardiac thrombus) accept Direct-Current Cardioversion within one week. anticoagulation (INR 2.0 to 3.0) is recommended for at least 3 weeks prior to and 4 weeks after cardioversion.
  Other Names: Cardioversion
  Arms: renal sympathetic denervation

SUMMARY:
To study whether renal sympathetic denervation(RSD) is safe and effective in patients with drug-resistant hypertension and symptomatic atrial fibrillation.

DETAILED DESCRIPTION:
Atrial fibrillation(AF) is the most common arrhythmia, and its frequency increases with age. Hemodynamic impairment and thromboembolic events related to AF result in significant morbidity, mortality, and cost. Management of patients with AF involves 3 objectives-correction of the rhythm disturbance, rate control, and prevention of thromboembolism. Regardless of whether the rate-control or rhythm-control strategy is pursued, attention must also be directed to antithrombotic therapy for prevention of thromboembolism. Pharmacological cardioversion approaches appear simple but are less efficacious. The major risk is related to poor tolerance of side effects，drug-associated toxicity，and proarrhythmic potentia1 of antiarrhythmic drugs. Radiofrequency catheter ablation of AF has developed rapidly in recent years, but the number of AF recurrences during the long-term follow-up was significant. In addition, the complications associated with AF ablation procedures likely to result in prolonged hospitalization, long-term disability or death. Hypertension is the most important risk factor for AF , Hypertension is associated with left ventricular hypertrophy, impaired ventricular filling, left atrial enlargement, and slowing of atrial conduction velocity. These changes in cardiac structure and physiology favor the development and maintenance of AF, and they increase the risk of thromboembolic complications. In patients with AF, aggressive treatment of hypertension may reverse the structural changes in the heart, reduce thromboembolic complications, and retard or prevent the occurrence of AF. Recently, many clinical researches have verified that Catheter-based renal sympathetic denervation can safely be used to substantially reduce blood pressure, reduce left ventricular hypertrophy, improve glucose tolerance and sleep apnea severity. Simultaneously, a marked reduction in muscle and whole-body sympathetic-nerve activity(MSNA) is apparent, with a decrease in renal and whole-body norepinephrine spillover. Left ventricle hypertrophy, left atrial enlargement, high norepinephrine level，glucose tolerance abnormity and obstructive sleep apnea are all recognized as independent risk factors for the development and recurrence of AF. So, we design this randomized parallel control multi center clinical study to demonstrate whether renal sympathetic denervation is safe and effective in patients with hypertension and symptomatic atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. Individual is ≥18 and ≤75 years of age
2. More than half a year for definite primary hypertension
3. Individual has a systolic blood pressure ≥160 mmHg (≥150 mmHg for type 2 diabetics) based on an average of three office blood pressure readings measured
4. Individual is adhering to a stable drug regimen, including three or more antihypertensive medications of which one is a diuretic, for a minimum of 14 days prior to enrollment
5. At least 30 seconds on a rhythm strip in an ECG record and at least 1 AF outbreak which was recorded by EGG and Holter during the preceding 6 months
6. Paroxysmal and persistent AF individual
7. Agree to attend experimental clinic and sign written informed consent

Exclusion Criteria:

1. Secondary and white-coat hypertension
2. Permanent AF individual
3. Thrombus in left atrial appendage found by transesophageal echocardiography
4. Individual with severely enlarged left atria ≥55 mm
5. Individual has experienced renal artery stenosis, or a history of prior renal artery intervention including balloon angioplasty or stenting, or ineligible conditions seen on renal artery computed tomography angiogram inspection such as double renal artery on one side, renal artery length ≤2 cm, diameter ≤4 mm, and distortion at incept sect
6. Individual has experienced a definite acute coronary syndrome in the past 3 months, or a cerebrovascular accident and alimentary canal bleeding within 3 months
7. Individual has experienced sick sinus syndrome
8. reversible causes of AF, including alcohol abuse, surgery, electrocution, myocadial infarction, pericarditis, myocarditis, pulmonary embolism or other pulmonary diseases, hyperthyroidism, and other metabolic disorders
9. structural heart diseases such as congenital, valvular heart diseases and kinds of cardiomyopathy
10. Individual is pregnant or nursing
11. Mental disorders - individual cannot complete follow-up or one the researcher thinks is unfit to be included in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-10 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Change in atrial fibrillation burden | from Baseline and 12 months
  to demonstrate the effect of RSD on AF burden in patients with drug-resistant hypertension and symptomatic AF.

SECONDARY OUTCOMES:
rate controlling in persistent AF patients | from baseline to 12 months
  to demonstrate the effect of RSD on rate controlling in persistent AF patients from baseline to 12 months post-randomization,
office systolic blood pressure | from baseline to 12 months
  the change in office systolic blood pressure from baseline to 12 months post-randomization
changes in cardiac structure and function,autonomic nerve function,fasting blood glucose, glycated hemoglobin, blood lipid, apnea-hypopnea index, pulse wave velocity and quality of life | from baseline to 12 months
  changes in cardiac structure and function by echocardiogram (include left ventricular ejection fraction, left ventricular end-diastolic diameter, interventricular septum, left atrium diameter), autonomic nerve function (heart rate variability by Holter), fasting blood glucose, glycated hemoglobin, blood lipid, apnea-hypopnea index, pulse wave velocity and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Qijun Shan, professor, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Qiu M, Yin Y, Shan Q. Renal sympathetic denervation versus antiarrhythmic drugs for drug-resistant hypertension and symptomatic atrial fibrillation (RSDforAF) trial: study protocol for a randomized controlled trial. Trials. 2013 Jun 11;14:168. doi: 10.1186/1745-6215-14-168. PMID 23759000